CLINICAL TRIAL: NCT07316699
Title: Evaluation of the Psychometric Properties of the Turkish Version of the Hypoglycaemia Self-Care Behaviour Scale
Status: Not yet recruiting | Type: Observational
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Principal Investigator, Semanur Bilgiç, research assistant, Bilecik Seyh Edebali Universitesi
Other Study IDs: semanur bilgiç diyabet ölçek
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus (DM); Hypoglycaemia; Self Care
Keywords: diabetes mellitus; Hypoglycaemia; Self-Care Behaviour; Scale
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to validate the validity and reliability of the Hypoglycaemia Self-Care Behaviour Scale, developed to assess hypoglycaemia self-care behaviours in patients with type 2 diabetes, through a prospective cross-sectional study.

DETAILED DESCRIPTION:
Diabetes is a chronic metabolic disease with a rapidly increasing prevalence worldwide that significantly impacts individuals' quality of life. One of the primary goals in diabetes management is to maintain optimal glycaemic control in order to prevent both acute and chronic complications. However, hypoglycaemia, which occurs when blood glucose levels drop to dangerous levels, particularly in individuals using insulin or sulphonylurea group drugs, is not only a significant clinical problem but also a powerful source of psychological stress. As an acute complication of diabetes, hypoglycaemia can have serious consequences for the patient's health. Therefore, the management and prevention of hypoglycaemic events are very important in diabetes self-care.

People with diabetes need comprehensive knowledge and self-care skills, including regular blood glucose monitoring, diet, exercise, and medication management, to effectively self-manage their condition and achieve optimal glycaemic control. Only patients with the correct care information can demonstrate appropriate self-care behaviour.

The fact that individuals with diabetes face lifelong management challenges emphasises the importance of correct self-care behaviours. In this context, rapid assessment tools are needed to evaluate behaviours for coping with and preventing hypoglycaemic episodes. The aim of this study is to validate the validity and reliability of the Hypoglycaemia Self-Care Behaviour Scale, developed to assess hypoglycaemia self-care behaviour in diabetic patients, in the Turkish population.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older,
* With type 2 diabetes mellitus,
* Who have had blood sugar levels <70 mg/dL at least once in the last six months,
* Who can read and write Turkish and communicate effectively.

Exclusion Criteria:

* Patients diagnosed with mental and/or cognitive disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetes patients receiving outpatient treatment under follow-up at the diabetes clinic
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Hypoglycaemia Self-Care Behaviour Scale | 6 months
  Developed in 2025 by Huang and colleagues. The scale consists of 10 items and 4 subscales: 'recognising hypoglycaemia and carbohydrate supplementation', 'preventing hypoglycaemia during exercise', 'carbohydrate assessment' and 'seeking medical help'. Each item is rated on a 5-point scale ranging from 1 (never) to 5 (always). The maximum possible score on the scale is 50, and scores below 30 indicate a need for hypoglycaemia education. The internal consistency of the developed scale ranges from 0.73 to 0.94, indicating strong reliability (Huang et al., 2025).

SECONDARY OUTCOMES:
Hypoglycaemic Confidence Scale | 6 months
  A 9-item self-report scale developed in 2017 by William Polonsky et al. to examine the degree to which people with diabetes feel confident and comfortable in their ability to protect themselves from hypoglycaemic problems. It was adapted into Turkish in 2021 by Büyükkaya Besen and Dervisoglu. Scale items are scored on a 1-4 scale. The ninth scale item for individuals with diabetes who have a partner is interpreted as follows: 1; does not trust at all 2; trusts a little 3; trusts moderately 4; trusts a lot. Scale scores are calculated by dividing the total item score by the number of completed items (for participants without a spouse, the calculation is based on 8 items).It is a unidimensional measure; an increase in the average score obtained from the scale indicates an increase in the level of confidence. The scale has no cut-off point.